CLINICAL TRIAL: NCT00912756
Title: Evaluation of Antiplatelet Therapy in Lower Limb Endovascular Treatment
Brief Title: Sufficient Treatment of Peripheral Intervention by Cilostazol
Acronym: STOP-IC
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kansai Rosai Hospital (Other)
Collaborators: Association for Establishment of Ebvidence in Interventions (Unknown)
Responsible Party: Osamu Iida, Kansai Rosai Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: STOP-IC
Record Dates: First submitted 2009-06-02; First posted 2009-06-03 (Estimated); Last update posted 2010-07-22 (Estimated); Status verified 2010-07

CONDITIONS: Arteriosclerosis Obliterans
Keywords: endovascular therapy; restenosis; cilostazol; femoropopliteal artery lesions; Chronic arteriosclerosis obliterans afflicting the femoropopliteal artery area
MeSH Terms: conditions — Arteriosclerosis Obliterans | interventions — Cilostazol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1cilostazol (Experimental): Cilostazol group: Treatment with cilostazol 200 mg/day BID (morning and evening) and aspirin at 100 mg/day will be started 3 to 7 days prior to EVT and continued until the end of the 2-year follow-up period.
  Interventions: Drug: cilostazol
- 2aspirin (Active Comparator): Non-cilostazol group: Treatment with aspirin 100 mg/day will be started 3 to 7 days prior to EVT and continued until the end of the 2-year follow-up period.
  Interventions: Drug: cilostazol

INTERVENTIONS:
Drug: cilostazol — 200 mg/day BID

SUMMARY:
Recently, Nanto et al. reported that cilostazol effectively prevented restenosis in a retrospective analysis of 121 femoropopliteal artery lesions in percutaneous transluminal angioplasty (PTA) patients who had undergone PTA. In a prospective 3-year follow-up study in 127 patients with similar diseases, the patency rate was significantly higher in the cilostazol group than in the ticlopidine group. It was also found that cilostazol markedly inhibited restenosis during the first 1-year period following endovascular therapy when restenosis is most frequently observed. In addition, there have been sporadic reports that cilostazol was effective in preventing post-stenting restenosis in the coronary artery area.

Based on these results, this multicenter study is going to be conducted to prospectively evaluate the usefulness of cilostazol in lower limb endovascular therapy.

ELIGIBILITY:
Patient criteria:

* Chronic arteriosclerosis obliterans afflicting the femoropopliteal artery area*
* Patients who can be monitored for at least 2 years after surgery

Lesion criteria:

* Angiographically-confirmed new significant superficial femoral artery stenosis or occlusive lesions that are 30 cm long or less if stented
* At least 1 arterial runoff below the knee; stenosis lesions not limiting flow may be included.
* Occlusive lesions may be included.

Exclusion criteria:

* Patients with or at risk of hemorrhagic complications or patients with bleeding tendency
* Patients with congestive cardiac failure
* Patients with a drug-eluting stent
* Patients with acute lower limb ischemia
* Patients with creatinine of 2 mg/dL or more(without dialysis)
* patients with a history of serious adverse reaction such as leukopenia, hepatic dysfunction, or renal dysfunction, or hypersensitivity to any component of the study drug.

Lesion criteria:

* Remnant inflow
* Severe calcification
* No arterial runoff below the knee

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2009-03; Primary Completion 2012-06 (Estimated); Study Completion 2012-09 (Estimated)

PRIMARY OUTCOMES:
Angiographic restenosis rate | 12 months +- 1 month

SECONDARY OUTCOMES:
Cardiovascular events

CONTACTS AND LOCATIONS:
Overall Officials: Osamu Iida, Study Director — Kansai Rosai Hospital
Locations (13):
- Japan (13):
  - Shinkoga Hospital, Kurume, Fukuoka
  - Hyogo College of Medicine Hopital, Nishinomiya, Hyōgo
  - Department of Cardiology, Kanazawa Cardiovascular Hospital, Kanazawa, Ishikawa-ken
  - Department of Cardiology,Naganoken Koseiren Shinonoi, Nagano, Nagano
  - Omihachiman Community Medical Center, Ōmihachiman, Shiga
  - Kansai Rosai Hospital and seven others, Amagasaki
  - Kishiwada Tokushukai Hospital, Kishiwada
  - Kokura Memorial Hospital, Kitakyusy
  - Shinshu University Hospital, Matsumoto
  - Caress Sapporo Tokeidai Memorial Hospital, Sapporo
  - Sendai Kousei Hospital, Sendai
  - Kikuna Memorial Hospital, Yokohama
  - Saiseikai Yokohama- City Eastern Hospital, Yokohama

REFERENCES:
- [Derived] Soga Y, Hamasaki T, Edahiro R, Iida O, Inoue N, Suzuki K, Yokoi Y, Kawasaki D, Zen K, Urasawa K, Aodo K; STOP-IC investigators. Sustained Effectiveness of Cilostazol After Endovascular Treatment of Femoropopliteal Lesions: Midterm Follow-up From the Sufficient Treatment of Peripheral Intervention by Cilostazol (STOP-IC) Study. J Endovasc Ther. 2018 Jun;25(3):306-312. doi: 10.1177/1526602818771358. Epub 2018 Apr 30. PMID 29706129
- [Derived] Iida O, Yokoi H, Soga Y, Inoue N, Suzuki K, Yokoi Y, Kawasaki D, Zen K, Urasawa K, Shintani Y, Miyamoto A, Hirano K, Miyashita Y, Tsuchiya T, Shinozaki N, Nakamura M, Isshiki T, Hamasaki T, Nanto S; STOP-IC investigators. Cilostazol reduces angiographic restenosis after endovascular therapy for femoropopliteal lesions in the Sufficient Treatment of Peripheral Intervention by Cilostazol study. Circulation. 2013 Jun 11;127(23):2307-15. doi: 10.1161/CIRCULATIONAHA.112.000711. Epub 2013 May 7. PMID 23652861